CLINICAL TRIAL: NCT01448538
Title: Non-Persistence/Non-Adherence of German wAMD Patients Related to Their Anti-VEGF Injections: Extent, Explanations and Patients' Preferences
Brief Title: Non-Persistence/Non-Adherence (NP/NA) in Wet Age-related Macular Degeneration (wAMD) Patients in Germany
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15785; HE-WAMD-01 (Other: Company internal)
Record Dates: First submitted 2011-10-04; First posted 2011-10-07 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Wet Macular Degeneration
Keywords: Medication Non-Adherence; Medication Persistence; wet macular degeneration
MeSH Terms: conditions — Wet Macular Degeneration; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Anti-VEGF injections

INTERVENTIONS:
Drug: Anti-VEGF injections — All Anti-VEGF injections approved for the German market, dosages as defined by doctors

SUMMARY:
In the research study an observation of patients with wet age-related macular degeneration (wet AMD) will be performed.

The term observational study indicates that the current course of therapy and the associated circumstances will be recorded. In this study, no medical care is changed. Also, no new drugs are tested.

This study is being conducted in about 30 centers in Germany. A total of approximately 500 patients will be enrolled. The study is designed for a period of 12 months.

At the beginning and end of the study the physician will document the patient data. Therefore will be used information from the patient records and documented visits. If such information is not available in the study center, the otherwise attending ophthalmologist will be consulted about the vision acuity values and visits in the observation period.

Furthermore, patients are asked to participate in three telephone interviews and fill out during their visits to the study center a short questionnaire about their current vision and their well-being. In the telephone interviews will be discussed with the patient about his wet AMD disease and its treatment, its experience and its perspectives as well as any problems occur.

ELIGIBILITY:
Inclusion Criteria:

* Patient has wet age-related macular degeneration (wAMD)
* Patient has already received at least one Anti-VEGF injection
* From a clinical standpoint, if there is an ophthalmological need for treatment it is probable that the patient gets additional anti-VEGF injections in the next year.
* The patient is able and willing to take part in the study (answering a short questionnaire in the study centre, 4 independent phone interviews during study period).

Exclusion Criteria:

* At time of inclusion visit, the study centre is only exceptionally responsible for the treatment of the patient.
* The patient is taking part in another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: German wAMD patients with Anti-VEGF therapy included by centers responsible for intravitreal injections
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2011-08; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Non-Persistence (NP) in the wAMD therapy in alternative study-specific definitions: (1) no eye exam for a period of at least 3 months OR (2) no 2 subsequent Anti-VEGF injections despite a clear medical need for injections | 12 months after a patient was included into the study

SECONDARY OUTCOMES:
Extent of Non-Adherence (NA) in the Anti-VEGF-therapy in a study-specific definition: (1) no eye exam every 4th week OR (2) no Anti-VEGF injection despite a medical need for an injection | 12 months after inclusion of patients
Identifying NA/NP causes (multivariate analysis based on patient interviews; main factors are sociodemographics and patient preferences) | Measurement during patient interviews about 4/8 months after inclusion
Identifying NA/NP outcomes (assessed by visual acuity) | Every eye doctors visit between inclusion of patients and their exclusion
Identifying patients' preferences (based on patients' questionnaires) towards treatment and treatment schemes | Measurement during patient interview after about 11 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Germany